CLINICAL TRIAL: NCT03375060
Title: Optimizing Patient Outcomes Through Early Detection of Uncontrolled Acid Reflux After Endoscopic Therapy in Barrett's Esophagus
Brief Title: Histology Post-Endoscopic Eradication Therapy (EET)
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Sponsor
Other Study IDs: STU00205592
Record Dates: First submitted 2017-10-16; First posted 2017-12-15 (Actual); Last update posted 2017-12-15 (Actual); Status verified 2017-12

CONDITIONS: Esophageal Reflux; Barrett Esophagus
MeSH Terms: conditions — Gastroesophageal Reflux; Barrett Esophagus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is looking at a cohort of patients who have undergone treatment for Barrett's Esophagus (BE) and who have experienced complete eradication of the disease. The aim of the proposed study is to evaluate the histologic features of the neosquamous epithelium (NSE) following complete eradication of intestinal metaplasia (CE-IM) in patients undergoing routine surveillance biopsies and compare these data to a direct measure of reflux using 24hr pH impedance, to determine the correlation between histology and persistent reflux. These data will allow us to more accurately risk stratify patients for recurrence of BE following EET.

ELIGIBILITY:
Inclusion Criteria:

* - Patients who have undergone endoscopic eradication therapy and 24hr pH impedance testing as part of standard of care between 2009 and 2014.
* - Individuals who have signed a consent to be part of the Prospective Evaluation of Barrett's Esophagus Study population.

Exclusion Criteria:

* - Individuals who are not yet adults (infants, children and teenagers), pregnant women and prisoners will be excluded from the study.
* - Patient who were previously unable or unwilling to give consent to the Prospective Evaluation of Barrett's Esophagus Study will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone EET and 24hr pH impedance testing as part of standard of care at Northwestern Memorial Hospital between 1/1/2009 and 12/31/2014 and who have enrolled in the Prospective Evaluation of Barrett's Esophagus database (NCT02634645).
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2017-11-05 (Actual); Study Completion 2017-11-05 (Actual)

PRIMARY OUTCOMES:
Composite histologic score of neosquamous epithelium following endoscopic eradication therapy (EET) | 1 year
  A composite histologic score made up of the following criteria:
  * Eosinophil infiltration (0: none, 1: scattered or focal, 2: diffuse or multifocal)
  * Dilated intercellular spaces (0: none, 0.5: intercellular spaces seen at 40x focal, 1: intercellular spaces seen at 40x diffuse, 1.5: intercellular spaces seen at 10x focal, 2: intercellular spaces seen at 10x diffuse)
  * Parakaratosis (0: absent, 2: present)
  * Ballooning degeneration (0: none, 1: focal, 2: extensive)
  * Basal cell hyperplasia (0: <15% of total thickness, 1: 15-33% of total thickness, 1.5: 33-66% of total thickness, 2: >66% of total thickness)
  * Columnar differentiation (0: no columnar mucosa present, 2: columnar mucosa adjacent to squamous)
  * Ulceration/erosion (0: absent, 1: present)
  Total possible score: 13

SECONDARY OUTCOMES:
24hr pH-impedance testing: percent acid reflux | 1 year
  Percent acid reflux
24hr pH-impedance testing: baseline impedance | 1 year
  Baseline impedance
24hr pH-impedance testing: Demeester score | 1 year
  Demeester score
Correlation between histologic features and persistent reflux | 1 year
  If participants with abnormal 24hr pH-impedance testing, as determined by outcomes 2, 3, and 4, have greater mean scores for histologic criteria evaluated in outcome 1.
Recurrence rate of intestinal metaplasia (Barrett's esophagus) | 1 year
  Recurrence rate of intestinal metaplasia in the overall cohort and the cohort with abnormal 24hr pH-impedance testing

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No